CLINICAL TRIAL: NCT01535664
Title: An Open-label, Proof of Concept Study to Evaluate Multiple Gait and Balance Parameters After Withdrawal of Dalfampridine-ER 10mg in Subjects With MS
Brief Title: An Open Label, Proof of Concept Study to Evaluate the Effects of Dalfampridine Withdrawal on Gait and Balance Parameters in Subjects With Multiple Sclerosis (MS)
Status: Completed | Type: Observational
Sponsor: Acorda Therapeutics (Industry)
Collaborators: Prometrika, LLC (Industry); BCS Consulting, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMP-MS-1008
Record Dates: First submitted 2012-02-07; First posted 2012-02-20 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dalfampridine-ER 10mg: Subjects with MS taking dalfampridine-ER 10mg and considered to be responders
  Interventions: Other: Withdrawal of dalfampridine-ER 10mg

INTERVENTIONS:
Other: Withdrawal of dalfampridine-ER 10mg — Withdrawal of dalfampridine-ER 10mg (7 days on study drug followed by withdrawal period of 10 days, followed by on study drug until study completion)
  * On drug Day-7 (visit 1) through Day 1 (visit 2)
  * Off drug Day 5±2 days (visit 3) through Day 11±2 days (visit 4)
  * On drug Day 15±2 days (visit 5)
  Other Names: Ampyra®

SUMMARY:
The purpose of this study is to determine changes on overall gait as well as in multiple gait and balance parameters after withdrawal of dalfampridine-ER 10mg in MS subjects who are receiving the medication consistently for at least two weeks prior to screening.

DETAILED DESCRIPTION:
Longitudinal study design

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* Receiving Ampyra® consistently for at least 2 weeks prior to the screening visit
* No history of seizures except simple febrile seizures

Exclusion Criteria:

* Sexually active woman of childbearing potential who is not surgically sterile, <two years post-menopause or is not using effective birth control methods
* Subject who is pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS Population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Pardo, MD, Principal Investigator — OMRF Multiple Sclerosis Center of Excellence
Locations (1):
- OMRF Multiple Sclerosis Center of Excellence, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalfampridine-ER 10mg: Subjects with MS taking dalfampridine-ER 10mg and considered to be responders
  Withdrawal of dalfampridine-ER 10mg : Withdrawal of dalfampridine-ER 10mg (7 days on study drug followed by withdrawal period of 10 days, followed by on study drug until study completion)
Period: Overall Study
Arm/Group | Dalfampridine-ER 10mg
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dalfampridine-ER 10mg
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Composite Score Overall Gait After Withdrawal and Reinitiation of Dalfampridine-ER 10mg
Description: The co-primary efficacy variable was overall gait. This novel composite score was created from standardized individual NeuroCom test results (Z-scores).
  ZGAIT (Z-Score Gait) is the average of Walk Across (WA) measuring step width, step length, speed; Tandem Walk (TW) measuring step width, speed and end sway, and Step/Quick turn (SQT) measuring turn time and turn sway).
  Overall gait was calculated by transforming ZGAIT into a percentile using the standard normal distribution. This rescales the Z-score to a scale from 0 to 100. A higher score is indicative of better performance.
Time Frame: 11 days on drug (day-7 to day 1 + day 11 to day 15) and 10 days withdrawn (day 1 to day 11)
Population: Full Analysis Population (FAP)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Dalfampridine-ER Withdrawn: Subjects with MS taking dalfampridine-ER 10mg and considered to be responders
  Withdrawal of dalfampridine-ER 10mg : Withdrawal of dalfampridine-ER 10mg (7 days on study drug followed by withdrawal period of 10 days, followed by on study drug until study completion)
Arm/Group | Dalfampridine-ER Withdrawn | Dalfampridine-ER 10 mg
Number analyzed (Participants) | 20 | 20
units on a scale | 46.01 (23.716) | 51.40 (21.582)
Statistical Analysis 1: Comparison: Dalfampridine-ER Withdrawn vs Dalfampridine-ER 10 mg; The co-primary efficacy variable was overall gait. This novel composite score was created from standardized individual NeuroCom test results (Z-scores). Overall gait was the average of WA, TW, and SQT; a higher score is indicative of better performance; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis — A step-down procedure using the primary statistical analysis was followed. If the p-value for the overall gait was less than 0.05, then overall balance was tested in the same manner. Otherwise, the testing procedure was stopped; P-value is based on a mixed model ANOVA with a fixed effect for treatment; Difference in least square means = 4.04, 95% CI 2-sided [0.87 to 7.20], Standard Error of Mean 1.51

2. Secondary Outcome: Change on the Berg's Balance Scale (BBS) After Withdrawal and Reinitiation of Dalfampridine-ER 10mg
Description: The BBS is a 14-item scale that evaluates subjects ability to sit, stand, reach, maintain single-leg stance, and turn. The scoring is rated from 0 (cannot perform task) to 4 (normal performance of task) for each of 14 items. The maximum possible score is 56 and the lowest 0. A higher total score is indicative of better performance.
Time Frame: 11 days on drug (day-7 to day 1 + day 11 to day 15) and 10 days withdrawn (day 1 to day 11)
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dalfampridine-ER Withdrawn | Dalfampridine-ER 10mg
Number analyzed (Participants) | 20 | 20
units on a scale | 45.7 (7.26) | 47.3 (6.71)
Statistical Analysis 1: Comparison: Dalfampridine-ER Withdrawn vs Dalfampridine-ER 10mg; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; P-value is based on a mixed model ANOVA with a fixed effect for treatment; Difference in least square means = 1.7, 95% CI 2-sided [0.7 to 2.8], Standard Error of Mean 0.5

3. Secondary Outcome: Change on the Two Minute Walk Test (2MWT) After Withdrawal and Reinitiation of Dalfampridine-ER 10mg
Description: Subjects will walk without assistance for 2 minutes and the distance will be measured and timed by the use of a stop watch.
  A larger walking distance is indicative of better performance.
Time Frame: 11 days on drug (day-7 to day 1 + day 11 to day 15) and 10 days withdrawn (day 1 to day 11)
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Dalfampridine-ER Withdrawn | Dalfampridine-ER 10mg
Number analyzed (Participants) | 20 | 20
Meters | 119.381 (35.9033) | 129.044 (28.8752)
Statistical Analysis 1: Comparison: Dalfampridine-ER Withdrawn vs Dalfampridine-ER 10mg; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; P-value is based on a mixed model ANOVA with a fixed effect for treatment; Difference in least square means = 7.729, 95% CI 2-sided [2.507 to 12.950], Standard Error of Mean 2.495

4. Secondary Outcome: Change on the Timed 25 Foot Walk Test (T25FW) After Withdrawal and Reinitiation of Dalfampridine-ER 10mg
Description: The T25FW test is a measure of ambulatory function that provides quantitative data and is used widely in the MS population
  A higher walking speed is indicative of better performance
Time Frame: 11 days on drug (day-7 to day 1 + day 11 to day 15) and 10 days withdrawn (day 1 to day 11)
Population: Full Analysis Population
Measure: Mean (Standard Deviation); unit: Feet per second (ft/s)
Arm/Group | Dalfampridine-ER Withdrawn | Dalfampridine-ER 10mg
Number analyzed (Participants) | 20 | 20
Feet per second (ft/s) | 3.42 (1.062) | 3.78 (0.901)
Statistical Analysis 1: Comparison: Dalfampridine-ER Withdrawn vs Dalfampridine-ER 10mg; Test type: Superiority or Other; p < .001, Mixed Models Analysis; P-value is based on a mixed model ANOVA with a fixed effect for treatment; Difference in least square means = 0.36, 95% CI 2-sided [0.19 to 0.54], Standard Error of Mean 0.08

5. Primary Outcome: Composite Score Overall Balance After Withdrawal and Reinitiation of Dalfampridine-ER 10mg
Description: The co-primary efficacy variable was overall balance. This novel composite score was created from standardized individual NeuroCom test results (Z-scores).
  Overall balance is a weighted average of Sensory Organization Test (SOT) fixed surface eyes open, fixed surface eyes closed, walls moving eyes open, surface moving eyes open, surface moving eyes closed, surface and walls moving eyes open; Limits of Stability Test (LOS) measuring reaction time, movement velocity, endpoint excursion, maximum excursion and directional control; and Adaptation Test (ADT) measuring the averaged, raw sway and center of force during rotational disturbances. ZBAL (Z-Score Balance)= (ZSOT*0.5) + (ZADT*0.2) + (ZLOS*0.3)
  Overall balance was calculated by transforming ZBAL into a percentile using the standard normal distribution. This rescales the Z-score to a scale from 0 to 100. A higher score is indicative of better performance.
Time Frame: 11 days on drug (day-7 to day 1 + day 11 to day 15) and 10 days withdrawn (day 1 to day 11)
Population: Full Analysis Population (FAP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dalfampridine-ER Withdrawn | Dalfampridine-ER 10mg
Number analyzed (Participants) | 20 | 20
units on a scale | 55.10 (27.150) | 54.98 (24.160)
Statistical Analysis 1: Comparison: Dalfampridine-ER Withdrawn vs Dalfampridine-ER 10mg; The co-primary efficacy variable was overall balance. This novel composite score was created from standardized individual NeuroCom test results (Z-scores). Overall balance was a weighted average of SOT, LOS, and ADT; Test type: Superiority or Other; p = 0.434, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; P-value is based on a mixed model ANOVA with a fixed effect for treatment; Difference in least square means = -2.38, 95% CI 2-sided [-8.60 to 3.84], Standard Error of Mean 2.97

ADVERSE EVENTS:
Time Frame: Screening Visit (day-7, Visit 1) through 30 days after the last dose of investigational product taken in Period 3 (day 15, visit 5).
Description: All summaries of AEs were based on treatment-emergent AEs (TEAE). TEAE was defined as an AE with date of onset (or worsening) that occurred on or after the Screening Visit (Visit 1) through 30 days after the last dose of investigational product taken in Period 3.
Groups:
- Dalfampridine-ER 10mg: Subjects with MS taking dalfampridine-ER 10mg
  Withdrawal of dalfampridine-ER 10mg : Withdrawal of dalfampridine-ER 10mg (7 days on study drug followed by withdrawal period of 10 days, followed by on study drug until study completion)
Arm/Group | Dalfampridine-ER 10mg | Dalfampridine-ER Withdrawn
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalfampridine-ER 10mg (N=20) | Dalfampridine-ER Withdrawn (N=20)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.